CLINICAL TRIAL: NCT02948530
Title: Measurement of Lung Elastance and Transpulmonary Pressure Using Two Different Methods (Lungbarometry)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stefan Lundin (Other)
Responsible Party: Sponsor-Investigator, Stefan Lundin, Professor, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Other Study IDs: LUA-74204
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Classically lung elastance and transpulmonary pressure are measured from the difference in tidal variations of airway pressure subtracted by tidal variations i esophagus pressure divided by the tidal volume. This requires the presence of a esophageal balloon catheter which is cumbersome and costly. In this study values obtained as described above are compared to values obtained with a new method in which a stepwise increase in positive endexpiratory pressure (PEEP) is performed with a size of the lung volume increase which corresponds to the tidal volume which the patient is ventilated with. The measurements are performed in sedated and mechanically ventilated patients in the intensive care unit.

DETAILED DESCRIPTION:
Classically lung elastance and transpulmonary pressure are measured from the difference in tidal variations of airway pressure subtracted by tidal variations in esophageal pressure divided by the tidal volume (Method 1). This requires the presence of a esophageal balloon catheter which is cumbersome and costly.

In this study values obtained as described in Method 1 above are compared to values obtained with a new method (Method 2) in which a PEEP-step is performed with a size of the lung volume increase which corresponds to the tidal volume which the patient is ventilated with. Measurements using Method 1 and 2 are performed in sedated and mechanically ventilated patients in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

Mechanically ventilated patients in the intensive care unit

Exclusion Criteria:

Patients with chronic obstrucive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sedated and mechanically ventilated patients in the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of lung elastance and transpulmonary pressure | Within one hour
  Comparison of a new versus the classical method for measurement of transpulmonary pressure

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lundin, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided